CLINICAL TRIAL: NCT00877279
Title: A Randomized,Blinded,Controlled,Multicenter Study of the Safety and Effectiveness of Dermal Filler, Belotero® Soft, After Superficial to Mid Dermal Implantation for Correction of Mild Facial Wrinkles Over 4 Weeks.
Brief Title: Multicenter Study of the Safety and Efficacy of Dermal Filler, Belotero® Soft
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MUS 90028-0717/1
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-10

CONDITIONS: Facial Wrinkles
Keywords: Facial wrinkles; Nasolabial folds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belotero® Soft (Experimental): Comparator will be given into the opposite side of the face that Belotero® Soft was administered for facial wrinkles, such as nasolabial folds.
  Interventions: Device: Belotero Soft
- CosmoDerm1 (Active Comparator)
  Interventions: Device: CosmoDerm1

INTERVENTIONS:
Device: CosmoDerm1 — CosmoDerm1 is a single use syringe, injected into the mid dermal layer.
  Arms: CosmoDerm1
Device: Belotero Soft — Dermal Filler
  Arms: Belotero® Soft

SUMMARY:
This study is to determine the safety and effectiveness of Belotero® Soft compared to active comparator in the correction of mild facial wrinkles, such as nasolabial folds.

DETAILED DESCRIPTION:
The purpose of the study is to see if Belotero® Soft is safe and effective for correction of mild facial wrinkles, such as nasolabial folds. The second objective of the study is to see if Belotero® Soft works better than the active comparator. Subjects will receive Belotero® Soft injection to one side of the face and the active comparator to the other side of the face.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have bilateral facial wrinkles, such as nasolabial folds

Exclusion Criteria:

* Other nasolabial fold correction within 6 months prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The severity of the facial wrinkle | 2 weeks and 4 weeks

SECONDARY OUTCOMES:
Investigator and subject assessments | 2 weeks and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rhoda Narins, MD, Principal Investigator — Dermatology Surgery and Laser Center
Locations (5):
- United States (5):
  - Skin Care & Laser Physicians of Beverly Hills, Los Angeles, California
  - Maas Clinic, San Francisco, California
  - Savin Dermatology Center, New Haven, Connecticut
  - William Coleman, III, MD, Metairie, Louisiana
  - Dermatology Surgery and Laser Center, White Plains, New York